CLINICAL TRIAL: NCT01762033
Title: A Multi-Center, Open-Label, Single-Arm, Phase 2 Study of ASONEP™ (Sonepcizumab/LT1009) Administered as a Single Agent to Subjects With Refractory Renal Cell Carcinoma
Brief Title: A Phase 2 Study of ASONEP™ to Treat Unresectable and Refractory Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Lpath, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT1009-Onc-002
Record Dates: First submitted 2012-12-17; First posted 2013-01-07 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Renal cell cancer; ASONEP; Sonepcizumab
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — sonepcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASONEP (Experimental): ASONEP will be administered by intravenous infusion over 90 minutes at 15 mg/kg once a week every 4 consecutive weeks per cycle
  Interventions: Drug: ASONEP

INTERVENTIONS:
Drug: ASONEP — Intravenous infusion
  Other Names: Sonepcizumab; LT1009

SUMMARY:
This Phase 2a study will investigate the efficacy, safety and tolerability of ASONEP™ (sonepcizumab/LT1009) when administered intravenously once a week, every 4 weeks (or cycle), to subjects with refractory renal cell carcinoma (RCC) until the disease progresses. Subjects who have failed 3 prior treatments for RCC including vascular endothelial growth factor (VEGF) and/or mammalian target of rapamycin (mTOR) inhibitors or who have tumors that cannot be surgically removed will be eligible for screening.

DETAILED DESCRIPTION:
LT1009-Onc-002 is a Phase 2a open-label, multi-center study designed to evaluate the efficacy and safety of ASONEP (sonepcizumab/LT1009) monotherapy in subjects with advanced, unresectable, refractory RCC who have previously failed up to 3 therapies, including VEGF and/or mTOR inhibitors. Two cohorts will be enrolled for a total of up to 39 subjects. Subjects will receive an intravenous (IV) infusion of ASONEP™ over 90 minutes at 24 mg/kg once a week and progression-free survival (PFS) will be assessed after 8 weeks of treatment. Cohort 1 will enroll approximately 22 subjects. A second cohort of up to 17 subjects will be enrolled if at least 12 out of 22 subjects from Cohort 1 demonstrated PFS at 8 weeks. Weekly dosing will take place from the date of randomization until the date of first documented progression or date of death from any cause, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced recurrent or metastatic RCC
* Histological or cytological confirmation of clear cell RCC - core tissue biopsy of either primary tumor or metastatic lesion with paraffin-embedded tissue specimens if no prior nephrectomy
* Measurable disease by RECIST 1.1
* Had one prior therapy for unresectable RCC with a VEGF/VEGFR targeted therapy (sunitinib, sorafenib, other VEGFR TKI or bevacizumab) - One prior treatment with an mTOR inhibitor (everolimus, temsirolimus or sirolimus) for unresectable disease permitted-Prior immunotherapy (immunomodulators such as cytokines, interleukins, vaccines, etc.) such as IL-2 also permitted
* Male or non-pregnant, non-nursing female
* Life expectancy ≥3 months
* ECOG performance status of 0, 1 or 2
* Must not be receiving any concurrent anticancer therapy
* Baseline CT or MRI scans of measurable disease sites by RECIST 1.1 performed within 2 weeks of Day 0 - For subjects with bone metastases, baseline bone scan performed within 4 weeks of study entry
* Adequate organ and immune function (within 7 days of Day 0):

Hemoglobin >9 g/dL-Absolute neutrophil count >1500 cells/uL without growth factors-Platelet count ≥100x10^9/L without transfusion-Serum creatinine <2.0x ULN or creatinine clearance >40 mL/min-Total bilirubin <1.5x ULN-AST/ALT <2.5x ULN (or <5.0x ULN if liver metastases present)-INR and aPTT <1.5x ULN

* Subject lesions for arterial spin labeling (ASL) MRI ≥2.5cm by CT imaging
* Must understand, be able and willing to fully comply with study procedures

Exclusion Criteria:

* Prior treatment with >3 VEGF pathway and/or mTOR inhibitors for RC cancer
* History of other CNS disease (spinal cord compression, or evidence of symptomatic brain or leptomeningeal carcinomatosis)
* Major surgery within 4 weeks of Day 0
* Radiation therapy within 4 weeks of baseline/infusion. Prior palliative radiation to metastatic lesions is acceptable if there is at least one measurable, non-radiated lesion
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring parenteral antibiotics on Day 0
* Known or suspected intolerance or hypersensitivity to study materials or any excipients
* Evidence of bowel obstruction because of theoretical possibility of GI perforation with an anti-angiogenesis agent
* Severe hemorrhage within 4 weeks of screening
* History of GI perforation
* History of non-healing wounds including ulcer or delayed bone fractures
* Prolonged QTc interval on baseline ECG (>450 msec for males or >470 msec for females), cardiac dysrhythmias including atrial fibrillation, torsade de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (<60 bpm), heart block (excluding 1st degree block, being PR interval prolongation only), congenital long QT syndrome or new ST segment elevation or depression or new Q wave on ECG
* Secondary malignancy within the last 5 years, except for adequately-treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer
* Previously enrolled in an sonepcizumab study or into this study and subsequently withdrawn
* History of alcohol or other substance abuse within the last year
* Use of corticosteroids or other immunosuppression (if taking systemic steroids [vs. topical], at least 4 weeks must have passed since the last dose)
* Growth factors within 1 week of screening
* Serious medical conditions that might be aggravated by treatment or limit compliance
* Cerebrovascular accident or transient ischemic attack, or pulmonary embolism within 6 months prior to screening
* Participation in another clinical trial
* Other severe or intercurrent acute or chronic medical or psychiatric condition or laboratory abnormality that may increase risk associated with study participation or study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 8 weeks
  The study will use a two-cohort design based on an 8-week PFS rate. Treatment will be considered promising if at least 12 out of the first 22 eligible subjects entered in the Cohort 1 of the study are progression free at Week 8. Enrollment of Cohort 2 will then proceed and be considered worthy of further evaluation if at least 25 out of 39 eligible subjects are progression free at Week 8. If no efficacy signal is observed after enrollment of 22 subjects in Cohort 1, the second cohort will not be enrolled and the clinical study may be stopped.

SECONDARY OUTCOMES:
Safety and Tolerability - Incidence and frequency of adverse events and serious adverse events | 8 weeks
  The incidence and frequency of adverse events and serious adverse events

OTHER OUTCOMES:
Pharmacokinetics Trough Concentrations | Pre-dose, weeks 1, 2, 4 of Cycle 1; pre-dose, weeks 2, 4 of Cycle 2
  Descriptive statistics (mean, median, standard deviation and coefficient of variation) will be used to summarize trough concentrations. For subjects testing positive for anti-drug antibodies (ADA) to ASONEP, the relationship between plasma ADA titers and ASONEP trough concentrations will be evaluated.
Tumor Response Rate | 8 weeks
  Imaging-based tumor assessments will be performed and response determined according to RECIST 1.1 criteria
Changes in Surrogate Markers | 8 weeks
  Blood samples will be drawn for lymphocyte, antibody, cytokine, VEGF and basic fibroblast growth factor (bFGF) analysis
Changes in Anti-drug Antibodies | 8 weeks
  Plasma samples will be evaluated for presence of ADA. If presence of ADA in plasma is confirmed, titers of anti-ASONEP will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hazel, Study Director — Lpath, Inc.
Locations (5):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Inverness, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, Nashville, Tennessee